CLINICAL TRIAL: NCT03487315
Title: Major Allergen in Wheat Anaphylaxis in Thai Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 842/2559(EC3)
Record Dates: First submitted 2017-08-31; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Wheat Allergy; Anaphylaxis Food; Anaphylaxis Exercise
MeSH Terms: conditions — Wheat Hypersensitivity; Exercise-Induced Allergies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- specific IgE (Experimental): Different level of specific IgE and immunoblot
  Interventions: Diagnostic Test: immunoblot

INTERVENTIONS:
Diagnostic Test: immunoblot — immunoblot

SUMMARY:
* To study Major allergen in Wheat anaphylaxis in Thai population
* To study and compare demographic data between group of wheat anaphylaxis

DETAILED DESCRIPTION:
Wheat is one of the most common causes in food-induced anaphylaxis and food dependent, exercised induced anaphylaxis. Gold standard for diagnose food allergy is double blind placebo control food challenge, but it is a high risk procedure. The accuracy of skin prick test and specific IgE assay showed unsatisfactory results. It might be explained by these tests may not detect all of the major allergens in wheat allergic patients. Previous studies showed that the major allergens of wheat dependent, exercised induced anaphylaxis are omega5 gliadin, followed by high molecular weight glutenin. For IgE-mediated wheat allergy, the major allergens varied among studies, including omega5 gliadin, glutenin, alpha/beta/gamma gliadin, and the water-soluble part of wheat allergens. There is no study to direct compare the major allergen between patients who have low wheat specific IgE and very high wheat specific IgE. Also, there is no data about the major allergens of wheat anaphylaxis in Thai population.

ELIGIBILITY:
Inclusion Criteria:

* Wheat anaphylaxis patient aged 1-60 years, who received treatment at division of allergy, department of Pediatrics and Medicine, Siriraj Hospital from 2001 to 2016

Exclusion Criteria:

* Loss follow up
* No consent form
* Celiac disease, Autoimmune disease was diagnosed

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Major allergen sensitized by Thai Patients with Wheat anaphylaxis | 1 hour
  To Identify major allergen (most component of protein that cause wheat allergy) between wheat anaphylaxis (low Specific IgE and high Specific IgE) and wheat dependent, exercise induced anaphylaxis by using immunoblot method (Electrophoresis). The results will be shown in electrophoresis gel and can identify in molecular weight (KDa) of protein which represent to major allergen of wheat protein.

CONTACTS AND LOCATIONS:
Overall Officials: Punchama Pacharn, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

REFERENCES:
- [Result] Nilsson N, Sjolander S, Baar A, Berthold M, Pahr S, Vrtala S, Valenta R, Morita E, Hedlin G, Borres MP, Nilsson C. Wheat allergy in children evaluated with challenge and IgE antibodies to wheat components. Pediatr Allergy Immunol. 2015 Mar;26(2):119-25. doi: 10.1111/pai.12334. PMID 25601168